CLINICAL TRIAL: NCT04892524
Title: Investigation Into the Identification, Management and Follow-up of Incidental Lung Nodules.
Brief Title: Virtual Management of Lung Nodules
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Southern Adelaide Local Health Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SALHNLungNodules
Record Dates: First submitted 2021-05-07; First posted 2021-05-19 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Pulmonary Nodule, Solitary; Pulmonary Nodule, Multiple
Keywords: Pulmonary nodule; Lung nodule; Solitary pulmonary nodule; Lung cancer; Virtual clinic
MeSH Terms: conditions — Solitary Pulmonary Nodule; Multiple Pulmonary Nodules; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual multidisciplinary review (Experimental): Participants in this arm will be reviewed in a virtual clinic by a multidisciplinary team
  Interventions: Other: Virtual multidisciplinary review
- Face-to-face review (No Intervention): Participants in this group will be reviewed in a face-to-face clinic

INTERVENTIONS:
Other: Virtual multidisciplinary review — The virtual multidisciplinary review involves participants being reviewed by a multi-disciplinary team of specialist doctors, nurses and radiologists in a virtual environment. The team will analyse radiologic scans and make a recommendations for any follow-up scans, procedures or appointments that may be required
  Arms: Virtual multidisciplinary review

SUMMARY:
This is a study to determine how a virtual model for the management of lung nodules compares to a face-to-face clinic for patient satisfaction, quality of life and cost.

DETAILED DESCRIPTION:
Initial Steps:

1. Individuals that have been referred to the Respiratory Outpatient Department of Flinders Medical Centre for management of a lung nodule will have their referral data screened by a doctor to determine that the referral meets criteria for management in the outpatient department and which category of follow-up is required (triaging process).
2. Eligible referrals will be provided to the study's research assistant who will contact the individual to discuss the study in detail and obtain consent to participate.
3. Individuals that have consented to participate are randomly assigned to either the 'virtual model' of lung nodule management (a), or the 'face-to-face model' of lung nodule management (b). Each participant has a 50% chance (1 in 2) of being assigned to either group.

   1. The 'virtual model' involves participants' CT scan(s) being reviewed by a multi-disciplinary team of specialist doctors, nurses and radiologists in a virtual environment. The team will analyse these scans and make a recommendation for any follow-up scans, procedures or appointments that may be required. The team will contact each participant with a phone-call. Participants primary care providers will also receive a letter describing the review and plan. Participants are not required to physically attend the hospital or outpatient department for this review to occur.
   2. The 'face-to-face model' involves a face-to-face appointment in the Respiratory outpatient clinic at Flinders Medical Centre, where a doctor will review participants' CT scan(s) and make a plan for any follow-up scans, procedures or appointments that may be required. Primary care providers will be informed of the outcome of this visit. Participants are required to physically attend the clinic appointment for this review.

All participants in this research study will be asked to complete an initial set of two questionnaires. The questionnaires include:

* Participant information questionnaire - collects personal information and contact details, as well as specific health-related, occupational and lifestyle information.
* Hospital Anxiety and Depression Scale (HADS)

Once participants have had their face-to-face appointment or virtual review, they will be asked to complete four questionnaires at a 1-month and 3-month interval. The questionnaires include:

* Hospital Anxiety and Depression Scale (HADS)
* Patient experience questionnaire
* Patient economic impact questionnaire
* Modified Visit-specific satisfaction instrument (VSQ-9)

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* At least 1 IPN identified on CT imaging measuring 4-30 mm in maximal diameter
* CT slice thickness of 3 mm or less

Exclusion Criteria:

* Previous diagnosis of lung cancer
* History of haemoptysis
* Unexplained weight loss > 7 kg in the preceding 12 months
* Past history of malignancy within 5 years (excluding non-melanoma skin cancer)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2021-04-19 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Cost | 6 months
  Economic cost to participants and our health service, measured by an investigator-derived questionnaire asking participants to describe time spent engaging in the their health care and any direct costs associated with visits. Economical modelling will also be applied to determine the staffing and resource costs associated with provision of care to participants in each arm.

SECONDARY OUTCOMES:
Participant satisfaction | 6 months
  Participant satisfaction, measured by the Visit-Specific Satisfaction Instrument (VSQ-9)
Anxiety | 6 months
  Participant anxiety as measure by the Hospital Anxiety and Depression Scale (HADS), which is a questionnaire containing seven items each for depression and anxiety subscales. Scoring for each item ranges from zero to three, with three denoting highest anxiety or depression level. A total subscale score of >8 points out of a possible 21 denotes considerable symptoms of anxiety or depression.

CONTACTS AND LOCATIONS:
Overall Officials: Anand Rose, Principal Investigator — Southern Adelaide Local Health Network
Locations (1):
- Flinders Medical Centre, Bedford Park, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No